CLINICAL TRIAL: NCT04451083
Title: Multiple-dose Study of FOY-305 in Japanese Healthy Adult Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FOY-305-02
Record Dates: First submitted 2020-06-21; First posted 2020-06-30 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — camostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FOY-305 (Experimental)
  Interventions: Drug: FOY-305

INTERVENTIONS:
Drug: FOY-305 — Multiple-dose of FOY-305 will be administered orally at 4 times/day.

SUMMARY:
To investigate safety, tolerability and pharmacokinetics in Japanese healthy adult male subjects when FOY-305 is administered as multiple-dose orally.

ELIGIBILITY:
Inclusion Criteria:

1. Japanese healthy adult male subjects
2. Age (at the time of informed consent): ≥18 yeas, ≤ 45 yeas
3. BMI (at the time of screening test): ≥18.5 kg/m2, <25.0 kg/m2

Exclusion Criteria:

1. Subjects who are on a treatment for or with a history of respiratory, cardiovascular, psychiatric, neurologic, gastrointestinal, immunologic, hepatic, renal, hematopoietic or endocrine and/or other disease.
2. Subjects with current or with a history of severe allergy to drugs or foods
3. Subjects with current or with a history of drug or alcohol abuse
4. Subjects with a history of hypersensitivity caused by ingredients of this drug

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-08-17 (Actual); Study Completion 2020-08-17 (Actual)

PRIMARY OUTCOMES:
Adverse events [Safety and Tolerability] | Up to 10 days
  Number of participants with adverse events as assessed by CTCAE v5.0
Vital sign [Safety and Tolerability] | Up to 10 days
  Summary statistics of blood pressure
Vital sign [Safety and Tolerability] | Up to 10 days
  Summary statistics of pulse rate
Vital sign [Safety and Tolerability] | Up to 10 days
  Summary statistics of SpO2
Body temperature [Safety and Tolerability] | Up to 10 days
  Summary statistics of body temperature
Body weight [Safety and Tolerability] | Up to 10 days
  Summary statistics of body weight
ECG parameter test [Safety and Tolerability] | Up to 10 days
  Summary statistics of ECG parameter test (Heart Rate)
ECG parameter test [Safety and Tolerability] | Up to 10 days
  Summary statistics of ECG parameter test (RR)
ECG parameter test [Safety and Tolerability] | Up to 10 days
  Summary statistics of ECG parameter test (PR)
ECG parameter test [Safety and Tolerability] | Up to 10 days
  Summary statistics of ECG parameter test (QRS)
ECG parameter test [Safety and Tolerability] | Up to 10 days
  Summary statistics of ECG parameter test (QT)
ECG parameter test [Safety and Tolerability] | Up to 10 days
  Summary statistics of ECG parameter test (QTcF)
Laboratory test [Safety and Tolerability] | Up to 10 days
  Summary statistics of laboratory test (hematologic test)
Laboratory test [Safety and Tolerability] | Up to 10 days
  Summary statistics of laboratory test (blood biochemistry test)
Laboratory test [Safety and Tolerability] | Up to 10 days
  Summary statistics of laboratory test (blood coagulation test)
Laboratory test [Safety and Tolerability] | Up to 10 days
  Summary statistics of laboratory test (urinalysis)

SECONDARY OUTCOMES:
Cmax of FOY-251 [Pharmacokinetic] | Up to 10 days
  Assessment of the Cmax of FOY-251 (Active metabolite of FOY-305)
Tmax of FOY-251 [Pharmacokinetic] | Up to 10 days
  Assessment of the Tmax of FOY-251 (Active metabolite of FOY-305)
AUC of FOY-251 [Pharmacokinetic] | Up to 10 days
  Assessment of the AUC4h of FOY-251 (Active metabolite of FOY-305)
AUC of FOY-251 [Pharmacokinetic] | Up to 10 day
  Assessment of the AUClast of FOY-251 (Active metabolite of FOY-305)
AUC of FOY-251 [Pharmacokinetic] | Up to 10 days
  Assessment of the AUCinf of FOY-251 (Active metabolite of FOY-305)
T1/2 of FOY-251 [Pharmacokinetic] | Up to 10 days
  Assessment of the T1/2 of FOY-251 (Active metabolite of FOY-305)
CL/F of FOY-251 [Pharmacokinetic] | Up to 10 days
  Assessment of the CL of FOY-251 (Active metabolite of FOY-305)

CONTACTS AND LOCATIONS:
Overall Officials: Susumu Nakade, Study Director — Ono Pharmaceutical Co. Ltd
Locations (1):
- Fukuoka Clinical Site 01, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: No